CLINICAL TRIAL: NCT02900092
Title: Treatment-Resistant Depression Augmentation Therapy With An Analog of the Neuroactive Steroid Allopregnanolone: A Pilot Study
Brief Title: Augmentation of Treatment-Resistant Depression With An Analog of the Neuroactive Steroid Allopregnanolone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Karen Klahr Miller, MD, Professor of Medicine, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016P001182
Record Dates: First submitted 2016-09-09; First posted 2016-09-14 (Estimated); Results first posted 2019-02-18 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Major Depressive Disorder
Keywords: postmenopausal; women; depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — ganaxolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ganaxolone (Experimental): Participants received ganaxolone
  Interventions: Drug: Ganaxolone

INTERVENTIONS:
Drug: Ganaxolone — Participants received ganaxolone

SUMMARY:
Major depressive disorder (MDD) is highly prevalent and nearly 70% of individuals with MDD do not respond to standard antidepressant therapies despite adequate dosing. An effective and well-tolerated antidepressant augmentation therapy would have important clinical and public health implications. Neuroactive steroid hormones are known to directly activate neurotransmitter receptors in the brain, and thus are potential candidates for augmentation therapies to enhance the effect of traditional antidepressants. The investigators hypothesize that administration of an allopregnanolone analog in women with treatment-resistant depression will improve depressive symptoms.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is highly prevalent and can have profoundly negative consequences on one's health, well-being and productivity. Women are twice as likely as men to experience depression during their lifetimes. In fact, it is reported that twelve million women in the U.S. each year will experience depression, and that one in eight women will experience a clinical depressive episode during their lifetimes. Additionally, nearly 70% of individuals with MDD do not respond to standard antidepressant therapies despite adequate dosing. Therefore, the identification of an effective and well tolerated antidepressant augmentation therapy would have important clinical and public health implications. Neuroactive steroid hormones are known to directly activate neurotransmitter receptors in the brain, and thus are potential candidates for augmentation therapies to enhance the effect of traditional antidepressants. Specifically, allopregnanolone, a steroid hormone derived from progesterone, is a potent positive modulator of GABA action at GABA-A receptors, which are known to have positive effects on mood symptoms. Data suggest that depression, chronic stress and posttraumatic stress disorder may be associated with low central nervous system allopregnanolone levels. The investigators propose to administer an oral allopregnanolone analog to 10 postmenopausal women with treatment-resistant depression as an add-on therapy to their current treatment for a period of 8 weeks followed by a 2-week taper. The investigators hypothesize that administration of the oral allopregnanolone analog in women with treatment-resistant depression will improve depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Female, age 50-75
2. Postmenopausal
3. Major Depressive Disorder
4. Currently treated with SSRI or SNRI at adequate dose

Exclusion Criteria:

1. Serious suicide or homicide risk
2. Unstable medical illness
3. Substance use disorder
4. Psychosis
5. Use of hormones (estrogens, androgens or related hormones)
6. History of hormone responsive cancer
7. Receiving strong CYP3A4 inducers or inhibitors or who intend to consume grapefruit products regularly during the study
8. Alanine aminotransferase (ALT) or creatinine > 3x upper limit of normal

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-01-12 (Actual); Study Completion 2018-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen K Miller, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dichtel LE, Nyer M, Dording C, Fisher LB, Cusin C, Shapero BG, Pedrelli P, Kimball AS, Rao EM, Mischoulon D, Fava M, Miller KK. Effects of Open-Label, Adjunctive Ganaxolone on Persistent Depression Despite Adequate Antidepressant Treatment in Postmenopausal Women: A Pilot Study. J Clin Psychiatry. 2020 Jun 9;81(4):19m12887. doi: 10.4088/JCP.19m12887. PMID 32558402

RESULTS

PARTICIPANT FLOW:
Groups:
- Ganaxolone Treatment Arm: Participants randomized to ganaxolone treatment
Period: Overall Study
Arm/Group | Ganaxolone Treatment Arm
Started | 10
Completed | 9
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Ganaxolone Treatment Arm: Participants received ganaxolone
Arm/Group | Ganaxolone Treatment Arm
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10
Montgomery-Asberg Depression Rating Scale (MADRS) [Mean (Standard Deviation); unit: units on a scale] — The MADRS is a diagnostic questionnaire that is used to measure the severity of depressive episodes in patients with mood disorders. The minimum and maximum values are 0 and 60, respectively, (higher scores are more severe)
  units on a scale | 24.4 (5.1)

OUTCOME MEASURES:

1. Primary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Description: The MADRS is a diagnostic questionnaire that is used to measure the severity of depressive episodes in patients with mood disorders. The minimum and maximum values are 0 and 60, respectively, (higher scores are more severe).
Time Frame: Week 8
Population: Ten subjects started the study. One subject dropped out (did not complete the 8-week study). Therefore, data from 9 subjects were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ganaxolone Treatment Arm
Number analyzed (Participants) | 9
units on a scale | 12.8 (2.9)

ADVERSE EVENTS:
Time Frame: 8 weeks
Groups:
- Ganaxolone Treatment Arm: Participants received ganaxolone treatment
Arm/Group | Ganaxolone Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 10/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ganaxolone Treatment Arm (N=10)
Sleepiness and fatigue (General disorders) | 10
Dizziness (General disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-05-14): https://cdn.clinicaltrials.gov/large-docs/92/NCT02900092/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-08): https://cdn.clinicaltrials.gov/large-docs/92/NCT02900092/SAP_001.pdf